CLINICAL TRIAL: NCT04704934
Title: A Phase 3, Multicenter, 2-Arm Randomized, Open-Label Study of Trastuzumab Deruxtecan in Subjects With HER2-Positive Metastatic and/or Unresectable Gastric or Gastro-Esophageal Junction (GEJ) Adenocarcinoma Subjects Who Have Progressed on or After a Trastuzumab-Containing Regimen (DESTINY-Gastric04)
Brief Title: Trastuzumab Deruxtecan for Subjects With HER2-Positive Gastric Cancer or Gastro-Esophageal Junction Adenocarcinoma After Progression on or After a Trastuzumab-Containing Regimen (DESTINY-Gastric04)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-U306; 2020-004559-34 (EudraCT Number)
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer, Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric Cancer, Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Trastuzumab deruxtecan; T-DXd; DS-8201a; Ramucirumab; Paclitaxel
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — trastuzumab deruxtecan; Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trastuzumab deruxtecan (Experimental): Participants who will be randomized to receive a 6.4 mg/kg intravenous (IV) dose of trastuzumab deruxtecan once every 3 weeks on Day 1 of each 21-day cycle.
  Interventions: Drug: Trastuzumab deruxtecan
- Ramucirumab + paclitaxel (Active Comparator): Participants who will be randomized to receive a 8 mg/kg IV dose of ramucirumab on Days 1 and 15 in combination with 80 mg/m^2 IV dose of paclitaxel on Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — 6.4 mg/kg IV infusion every 3 weeks on Day 1 of each 21-day cycle
  Other Names: T-DXd; DS-8201a; ENHERTU®
  Arms: Trastuzumab deruxtecan
Drug: Ramucirumab — 8 mg/kg IV infusion on Days 1 and 15 of a 28-day cycle
  Other Names: CYRAMZA®
  Arms: Ramucirumab + paclitaxel
Drug: Paclitaxel — 80 mg/m^2 IV infusion on Days 1, 8, and 15 of a 28-day cycle
  Arms: Ramucirumab + paclitaxel

SUMMARY:
This study will evaluate the efficacy and safety of trastuzumab deruxtecan (T-DXd) compared with ramucirumab and paclitaxel (Ram + PTX) in participants with HER2-positive gastric or gastro-esophageal junction (GEJ) adenocarcinoma who have progressed on or after a trastuzumab-containing regimen and have not received any additional systemic therapy.

DETAILED DESCRIPTION:
This study will assess the efficacy and safety of T-DXd compared with Ram + PTX in participants with HER2-positive (defined as immunohistochemistry [IHC] 3+ or IHC 2+/in situ hybridization [ISH]+) gastric or GEJ adenocarcinoma (based on [American Society of Clinical Oncology (ASCO) College of American Pathologists (CAP) guidelines who have progressed on or after a trastuzumab-containing regimen and have not received any additional systemic therapy. Participants will be randomized 1:1 to either T-DXd or Ram + PTX treatment. The primary objective will assess overall survival. Secondary objectives will further assess progression-free survival, objective response rate, duration of response, disease control rate, safety, pharmacokinetics, and immunogenicity of T-DXd.

ELIGIBILITY:
Inclusion Criteria:

* Adults (according to local regulation) and able to provide informed consent for study participation.
* Pathologically documented gastric and GEJ adenocarcinoma that has been previously treated in the metastatic setting (unresectable, locally advanced, or metastatic disease).
* Progression on or after first-line therapy with a trastuzumab or approved trastuzumab biosimilar-containing regimen. Note: Prior neoadjuvant or adjuvant therapy with a trastuzumab-containing regimen can be counted as a line of therapy if the subject progressed on or within 6 months of completing neoadjuvant or adjuvant therapy. Prior neoadjuvant or adjuvant therapy that does not include trastuzumab will not be counted as a line of therapy regardless of the progression status of the subject.
* Locally or centrally confirmed HER2-positive (IHC 3+ or IHC 2+ and evidence of HER2 amplification by ISH) as classified by ASCO-CAP on a tumor biopsy obtained after progression on or after a first-line trastuzumab or approved trastuzumab biosimilar-containing regimen.
* Eastern Cooperative Oncology Group performance status of 0 or 1 at Screening.
* Adequate bone marrow, renal, hepatic function, and blood clotting function within 14 days of randomization.

Exclusion Criteria:

* Use of anticancer therapy after trastuzumab-containing treatment
* Medical history of myocardial infarction (MI) within 6 months before randomization/enrollment, symptomatic congestive heart failure (New York Heart Association Class II to IV).
* Has a QT interval corrected by Fridericia's formula (QTcF) prolongation to >470 msec (female subjects) or >450 msec (male subjects) based on average of the Screening triplicate12-lead ECG.
* Has a history of (non-infectious) interstitial lung disease (ILD/pneumonitis) that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
* Any autoimmune, connective tissue or inflammatory disorders (eg, rheumatoid arthritis, Sjögren syndrome, sarcoidosis, etc.) where there is documented (or a suspicion of) pulmonary involvement at the time of Screening.
* Prior complete pneumonectomy.
* Spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
* Has multiple primary malignancies within 3 years, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, other solid tumors curatively treated.
* History of severe hypersensitivity reactions to either the T-DXd or inactive ingredients in T-DXd.
* History of severe hypersensitivity reactions to other monoclonal antibodies, including ramucirumab or to any of its excipients.
* Known allergy or hypersensitivity to paclitaxel or any components used in the paclitaxel preparation or other contraindication for taxane therapy.
* Current uncontrolled infection requiring antibiotics, antivirals, or antifungals or an unexplained fever >38.0°C during Screening visits or on the first scheduled day of dosing (at the discretion of the Investigator, participants with tumor fever may be enrolled), which in the Investigator's opinion might compromise the participant's participation in the study or affect the study outcome
* Clinically significant gastrointestinal disorder (eg, including hepatic disorders, bleeding, inflammation, occlusion, ileus, diarrhea Grade >1, jaundice, intestinal paralysis, malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, or partial bowel obstruction) in the opinion of Investigator
* Has history of receiving live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first exposure to study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival in Participants Who Were Administered Trastuzumab Deruxtecan Compared With Ramucirumab in Combination With Paclitaxel | Time from date of randomization until death (due to any cause), up to approximately 36 months
  Overall survival (OS) is defined as the time from date of randomization until death from any cause.

SECONDARY OUTCOMES:
Progression-free Survival in Participants Who Were Administered Trastuzumab Deruxtecan Compared With Ramucirumab in Combination With Paclitaxel | Time from date of randomization until first objective radiographic disease progression or death (due to any cause) whichever occurs first, up to approximately 36 months
  Progression-free survival (PFS) is defined as the time from date of randomization until first objective radiographic tumor progression or death from any cause, based on Investigator assessment.
Objective Response Rate in Participants Who Were Administered Trastuzumab Deruxtecan Compared With Ramucirumab in Combination With Paclitaxel | From start of treatment to date of documented disease progression, up to approximately 36 months
  Objective response rate (ORR) is defined as the proportion of participants who achieve a best response of complete response (CR) or partial response (PR) using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by Investigator.
Duration of Response in Participants Who Were Administered Trastuzumab Deruxtecan Compared With Ramucirumab in Combination With Paclitaxel | Time from initial response (CR or PR) to date of documented disease progression or death (due to any cause) whichever occurs first, up to approximately 36 months
  Duration of response (DoR) is defined time from the initial response (CR or PR) until documented tumor progression or death from any cause and based on Investigator assessment.
Disease Control Rate in Participants Who Were Administered Trastuzumab Deruxtecan Compared With Ramucirumab in Combination With Paclitaxel | From start of treatment to date of documented disease progression, up to approximately 36 months
  Disease control rate (DCR) is defined as the proportion of participants who achieved CR, PR, or stable disease (SD) for a minimum of 6 weeks during study treatment, based on Investigator assessment.
Incidence of Treatment-emergent Adverse Events (TEAE), Serious Adverse Events (SAE), Adverse Events of Special Interest (AESI), and Physical Examination Findings | From time subjects signs informed consent form up to 40 days after last study dose
  Adverse events will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0.
Serum Concentrations for Trastuzumab Deruxtecan, total anti-HER2 antibody, and Active Metabolite MAAA-1181a | Cycles 1-4 and subsequent cycles on Day 1 pre- and post-infusion (each cycle is 28 days)
Percentage of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) | Cycles 1, 2, and 4 on Day 1 pre-infusion, then every 4 cycles on Day 1 pre-infusion, 40 day follow up until death, withdrawal of consent, or lost to follow up whichever occurs first (each cycle is 28 days)
  The immunogenicity of trastuzumab deruxtecan will be assessed.
Percentage of Participants Who Have Treatment-emergent ADAs | Cycles 1, 2, and 4 on Day 1 pre-infusion, then every 4 cycles on Day 1 pre-infusion, 40 day follow up until death, withdrawal of consent, or lost to follow up whichever occurs first (each cycle is 28 days)
  The immunogenicity of trastuzumab deruxtecan will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (156):
- Argentina (4):
  - Instituto Medico Especializado Alexander Fleming, Colegiales, Buenos Aires F.D.
  - IONC Instituto Oncologico de Cordoba - Fundacion Richardet Longo, Nueva Cordoba, Córdoba Province
  - Exelsus, San Miguel de Tucumán, Tucumán Province
  - Fundacion Cenit, Buenos Aires
- Belgium (4):
  - UCL St. Luc, Brussels
  - Antwerp University Hospital, Edegem
  - Pôle Hospitalier Jolimont, Haine-Saint-Paul
  - UZ Leuven, Leuven
- Brazil (4):
  - PERSONAL - Oncologia de Precisao e Personalizada, Belo Horizonte
  - Hospital Sirio Libanes, Brasília
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia LTDA, Ijuí
  - Hospital Ernesto Dornelles, Porto Alegre
- Chile (3):
  - SIM Centro de Investigacion Clinica, Temuco, Cautin
  - Fundacion Arturo Lopez Perez, Santiago, Santiago Metropolitan
  - Clinica San Carlos de Apoquindo, Santiago, Santiago Metropolitan
- China (24):
  - Anhui Provincial Hospital, Heifi, Anhui
  - Fujian Medical University - Fujian Provincial Cancer Hospital, Fuzhou, Fuijan
  - Xiamen University - The First Affiliated Hospital, Xiamen, Fujian
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - 1Affiliated H of Sun Yat Sen U, Guangzhou, Guangdong
  - Hebei Medical Univ 4th Hosp, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhongnan univ Xiangya hosp, Changshan, Hunan
  - Jiangsu Province Hosp, Nanjing, Jiangsu
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - 1st Hosp of China Medical Univ, Shenyang, Liaoning
  - Shandong Cancer Hospital & Institute, Jinan, Shandong
  - Zhongshan Hosp Fudan Univ, Shanghai, Shanghai Municipality
  - Shanghai First People's Hosp, Shanghai, Shanghai Municipality
  - Xinjiang Medical University - Cancer Hospital, Ürümqi, Xinjiang
  - Zhejiang Medical University - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - Peking Univ 3rd Hosp, Beijing
  - The 1st Hospital of Jilin Univ, Changchun
  - Sir Run Run Shaw Hospital, Hangzhou
  - Linyi Cancer Hospital, Linyi
  - 1 Affiliated H of Nanchang U, Nanchang
  - Fudan University - Shanghai Cancer Center, Shanghai
- France (11):
  - CHU Besançon, Besançon
  - CHRU, Brest
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital de la Timone, Marseille
  - Institut de Recherche en Cancerologie de Montpellier IRCM, Montpellier
  - Hopital Saint Antoine, Paris
  - L Institut Mutualiste Montsouris, Paris
  - Hopital Europeen G. Pompidou, Paris
  - Pharmacie ICLN, Saint-Priest-en-Jarez
  - Gustave Roussy, étage -1., Villejuif
- Germany (8):
  - Charité-Unimedizin Berlin, Berlin
  - Uniklinikum Carl-Gustav-Carus, Dresden Sachsen
  - Evang. Klin. Essen-Mitte gGmbH, Essen
  - Ins. für klinische onk. Forschung, Frankfurt Am Main Hessen
  - Häm-Onk. Praxis Eppendorf, Hamburg
  - Asklepios Tumorzentrum Altona, Hamburg
  - Uni zu Koln-Unikl. Koln, Kln Nordrhein-westfalen
  - Universitares Krebszentrum, Leipzig
- Hong Kong (4):
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Chinese University of Hong Kong (CUHK) - Prince of Wales Hospital (PWH) - Vascular and Interventional Radiology Foundation (VIRF) Clinical Science Centre, Hong Kong
- Hungary (3):
  - Magyar Honvedseg Egeszs. K, Budapest
  - Debreceni Egyetem Klinikai, Debrecen
  - Tolna M. Balassa Janos Korhaz, Szekszárd
- Ireland (4):
  - Cork University Hospital, Cork
  - Tallaght University Hospital, Dublin
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
- Israel (3):
  - Soroka Univ Medical CTR, Be'er-Sheva Southern
  - Davidoff Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
- Italy (11):
  - AOU Pisana, Barone
  - IRCC-FPO Candiolo, Candiolo
  - AOU Mater Domini, Catanzaro
  - Istituto Europeo di Oncologia S.r.L Divisione di Oncologia Medica Gastrointestinale e Tumori Neuroendocrini, Milan
  - Ospedale Niguarda, Milan
  - San Raffaele Hospital, Milan
  - Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Aou Vanvitelli, Napoli
  - Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
- Japan (12):
  - Aichi Cancer Center Hospital, Nagoya, Aichia
  - National Cancer Center Hospital, Chūōku
  - Osaka International Cancer Institute, Chūōku
  - Gifu University Hospital, Gifu
  - National Cancer Center Hospital East, Kashiwa
  - Kobe City Medical Center General Hospital, Kobe
  - Kochi Health Sciences Center, Kochi
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Niigata Cancer Center Hospital, Niigata
  - Kindai University Hospital, Ōsaka-sayama
  - Osaka University Hospital, Suita
- Poland (2):
  - Sklodowska-Curie Inst Oncology, Warsaw
  - Uniwersytecki Szpital Kliniczny im.Mikulicza-Radeckiego, Wroclaw
- Portugal (3):
  - Hospital Sra da Oliveira, Creixomil E Mariz
  - Instituto Portugues De Oncologia Do Porto Francisco Gentil, E.P.E., Porto
  - C Hosp Tras Montes Alto Douro, Vila Real
- Romania (4):
  - S.C. Oncopremium-Team SRL, Baia Mare
  - Institutul Oncologic Prof. Dr. Alexandru Trestiorean Bucuresti IOB, Bucharest
  - S.C. Medisprof SRL, Cluj-Napoca
  - Centrul de Oncologie Sf. Nectarie, Craiova
- Russia (4):
  - SBIH Chelyabinsk Regional Clinical Centre of Oncology and Nuclear Medicine, Chelyabinsk
  - Private Medical Institution "Euromedservice", Saint Petersburg
  - City Clinical Oncology Dispensary, Saint Petersburg
  - Republican Clinical Oncology Dispensary, Ufa
- Singapore (2):
  - National Univ Cancer Inst SGP, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (10):
  - Kyungpook Nat Uni Chilgok Hos, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul Nati Univ Bundang Hosp, Seongnam
  - Korea Univ Anam Hosp, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Marys Hospital, Seoul
  - Chonbuk National University Hospital - Jeonbuk Regional Cancer Center, Seoul
- Spain (9):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - H. Gregorio Maranon, Madrid
  - Hosp Univ Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital de Navarra, Pamplona
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela
  - H. Clinico U. de Valencia, Valencia
- Taiwan (8):
  - KMUH, Kaohsiung City
  - CGMF-Kaohsiung Branch, Kaohsiung City
  - China Medical Univ Hosp, Taichung
  - National Cheng Kung Univ Hosp, Tainan
  - National Taiwan University Hospital NTUH, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hosp, Taipei
  - CGMF-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (4):
  - SBU Adana Sehir Hastanesi, Adana
  - Trakya Universitesi Balkan, Edirne
  - Suleyman Yalcin Seh. Hast., Istanbul
  - Inonu Uni. Turgut Ozal Tip, Malatya
- Ukraine (3):
  - National Cancer Institute, Kyiv
  - MedicalCenter ASKLEPION LLC, Kyiv
  - LLC "Oncolife", Zaporizhzhia
- United Kingdom (12):
  - University Hospitals Birmingham UHB NHS Foundation Trust - Queen Elizabeth Hospital Birmingham QEHB, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Velindre NHS Trust - Velindre Cancer Centre VCC, Cardiff
  - Ninewells Hospital, Dundee
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - UCLH Trust, London
  - Royal Marsden NHS, London
  - Christie Hospital, Manchester
  - University of Oxford, The Churchill Hospital, Oxford
  - Royal Marsden Sutton, Sutton
  - Leeds Teaching Hospitals NHS Trust, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Shitara K, Van Cutsem E, Gumus M, Lonardi S, de la Fouchardiere C, Coutzac C, Dekervel J, Hochhauser D, Shen L, Mansoor W, Liu B, Fornaro L, Ryu MH, Lee J, Faustino C, Metges JP, Tabernero J, Franke F, Janjigian YY, Souza F, Jukofsky L, Zhao Y, Kamio T, Zaanan A, Pietrantonio F; DESTINY-Gastric04 Trial Investigators. Trastuzumab Deruxtecan or Ramucirumab plus Paclitaxel in Gastric Cancer. N Engl J Med. 2025 Jul 24;393(4):336-348. doi: 10.1056/NEJMoa2503119. Epub 2025 May 31. PMID 40454632